CLINICAL TRIAL: NCT04921904
Title: Phase I/II Study of Abemaciclib + Ramucirumab in Metastatic Esophageal/Gastroesophageal Junction Carcinomas
Brief Title: Abemaciclib Plus Ramucirumab for Esophageal/Gastroesophageal Junction Ca
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020-055
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Esophageal Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — abemaciclib; Ramucirumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abemaciclib plus Ramucirumab (Experimental): Abemaciclib 150mg dose administered orally twice daily every day plus Ramucirumab dose 8mg/kg iv every 2 weeks until evidence of disease
  Interventions: Drug: Abemaciclib; Drug: Ramucirumab

INTERVENTIONS:
Drug: Abemaciclib — 150mg dose administered orally twice daily every day
Drug: Ramucirumab — 8mg/kg iv every 2 weeks until evidence of disease

SUMMARY:
CDK4/6 and Cyclin D1 are significantly expressed in approximately 80% of esophageal and gastroesophageal junction tumors suggesting that CDK4/6 inhibition may be a successful strategy in these chemotherapy and immunotherapy resistant diseases.

DETAILED DESCRIPTION:
This is a multicenter, open label, phase I/II safety study that will enroll 30 subjects with metastatic esophageal and gastroesophageal junction adenocarcinomas post first line systemic chemotherapy. Subjects will be treated with oral Abemaciclib 150 mg PO daily bid given with ramucirumab 8mg/kg every 2 weeks iv until evidence of disease progression or unacceptable toxicities.

A total of 30 subjects will be enrolled. The primary goal is to describe the safety profile of Abemaciclib in combination with Ramucirumab among all enrolled subjects.

If grade 3 or higher treatment-related adverse events occur in 20 subjects, the upper bound of 95% Wilson confidence interval for the adverse event rate would be below 81% (16.7% - 47.9%).

The safety analysis will be performed in all treated subjects. Adverse event data will be listed individually and graded according to the National Cancer Institute Common Terminology Criteria, version 4.03.

Summary statistics will include counts and proportions as well as rates with 95% confidence intervals. Toxicities will be reported as a tabulated table by type and grade.

Objective response rate is defined as the percentage of subjects who achieve an objective response by RECIST1.1 criteria (i.e. Complete response or Partial Response) to Abemaciclib in combination with Ramucirumab. We will estimate the objective response rate, along with the Wilson 95% confidence interval, for the population of subjects.

Overall survival will be defined as the time from study enrollment to death. This will be summarized using a Kaplan-Meier curve.

The proportion of subjects with grade 4 or higher treatment-related adverse events will be monitored continuously throughout the trial using a Bayesian stopping guideline. A Beta (1, 19) prior, representing a toxicity rate of 5%, slightly lower than the expected rate of 6%, was used in the development of our guidelines. The therapy will be re-evaluated if the posterior probability that the toxicity rate exceeds 10% is greater than 75%. Table 3 summarizes the stopping boundaries starting with the initial cohort of 3 subjects through the maximum sample size of 30 subjects.

The probability of triggering the stopping guidelines was assessed for a range of possible toxicity rates using simulations with 5000 replicates. The probability of stopping to re-evaluate was 1% if the true proportion with an unacceptable toxicity was 5%. In comparison, the probability of stopping early was 99.6% if the true proportion with an unacceptable toxicity was 40%

ELIGIBILITY:
Subjects must meet all eligibility criteria. The key inclusion and exclusion criteria are as follows:

Key Inclusion Criteria:

* All subjects must have metastatic esophageal or gastroesophageal junction carcinomas (adenocarcinoma only)
* ECOG performance status of 0 or 1
* Tumor tissue must be available for correlative studies - Either a formalin fixed paraffin block or a minimum of ten 5-micron tissue section's (slides) of tumor biopsy sample must be available for biomarker evaluation.
* Patients must have received at least one prior line of standard systemic therapy for recurrent or Stage IV disease, and that patients with HER2 overexpression have received an anti-HER2 drug.

Key Exclusion Criteria:

* Squamous cell carcinomas
* Mixed histology with small cell component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To describe the safety profile of Abemaciclib + Ramucirumab as assessed according to Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0). | 24 months

SECONDARY OUTCOMES:
To assess objective response rate | 24 months
To assess progression free survival | 24 months
To assess overall survival | 24 months
To determine the rate of stable disease at 3 months post targeted therapy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Kelly, MD, Principal Investigator — Charles A Sammons Cancer Center/Texas Oncology
Locations (1):
- Baylor University Medical Center, Charles A Sammons Cancer Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No